CLINICAL TRIAL: NCT06146491
Title: A COMPARISON OF ANALGESIC EFFICACY OF TRANSDERMAL DICLOFENAC AND ORAL COMBINATION OF PARACETAMOL AND IBUPROFEN IN POSTOPERATIVE PAIN MANAGEMENT FOLLOWING SURGICAL EXTRACTION OF MANDIBULAR THIRD MOLAR
Brief Title: A COMPARISON OF TRANSDERMAL DICLOFENAC AND ORAL COMBINATION OF PARACETAMOL AND IBUPROFEN IN POSTOPERATIVE PAIN MANAGEMENT FOLLOWING SURGICAL EXTRACTION OF MANDIBULAR THIRD MOLAR- A RANDOMISD CONTROLLED TRIALS.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Niroj Khanal, NIROJ KHANAL, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRC/2223/022
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Tablets; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drugs (Active Comparator): oral combination of paracetamol (500mg) - ibuprofen (400mg) will be given to group A. they are provided in tablet and prescribed at 8 hourly for three days
  Interventions: Drug: Oral tablet and transdermal patch
- Drug (Active Comparator): Transdermal diclofenac patch - 200mg for group B. Patch is applied on right hand in deltoid region , and ask the patient to change patch every 24 hourly.
  Interventions: Drug: Oral tablet and transdermal patch

INTERVENTIONS:
Drug: Oral tablet and transdermal patch — oral combination of paracetamol -500mg and ibuprofen - 400mg will be given to group A and transdermal diclofenac patch - 200 mg will be given to group B.

SUMMARY:
This is comparative interventional study, will be conducted in patient indicated for surgical extraction of mandibular third molar at the Department of Oral and Maxillofacial surgery, College of Dental Surgery, BPKIHS, Nepal. Verbal and written will be taken . Participants meeting inclusion criteria will be included in the study and will be divided in to two groups, group A (Oral combination of paracetamol-500mg and ibuprofen -400mg) and group B ( Transdermal diclofenac patch-200mg) using computer generated randamization. Extraction will be carried out using standard protocol. Aformention drugs will given to participants accordingly for management of post operative pain.Tramadol will be given to each patient as rescue analgesics and allowed to have if pain score exceeds 7.post operative instruction will be given carefully. Rescue phone number will be provided in case of emergency. Telephonic interview will be performed at 12, 24 and 72 hours post operatively and pain score using numeric rating scale will be recorded.Any adverse effects of drugs will be recorded. The data collected will be entered in Microsoft excel sheet. It will then be transferred into SPSS (Statistical Package for Social Sciences) for statistical analysis.

DETAILED DESCRIPTION:
Introduction:unpleasant sensory and emotional experience associated with, or resembling that associated with, actual or potential tissue damage" is the new definition of pain as per IASP 2020. Pain is one of the most commonly experienced symptoms in oral and maxillofacial surgery and as such is a major concern to the surgeon. One of the most important aspects of the practice of dentistry is the control or elimination of pain. Pain is one of the most common post-operative complication following surgical removal of mandibular third molar extraction. To ameliorate the pain we commonly prescribe NSAIDS like oral Paracetamol ,ibuprofen, oral diclofenac sodium etc. Non steroidal anti inflammatory drugs work well to relieve mild to moderate intense postoperative pain. Their mechanism of action depends on whether they inhibit cyclooxygenase-1 (COX-1), cyclooxygenase-2 (COX-2), or both, which are responsible for the synthesis of different prostaglandins found in pathological situations (COX-2 is more expressed in inflammatory conditions). NSAIDS can be administered in a variety of routes, including oral, par-enteral, inhalation as well as trans dermal. Through Oral route is the most common for the drugs delivery. Oral route carries the risk of first pass metabolism and loss of substantial quantities of the drug before it is absorbed systemically. Par-enteral administration of drugs can be extremely painful and sudden increase in drug concentration in the plasma could lead to certain adverse effects. Trans dermal patches offer several advantages over the oral route such as bypassing first pass metabolism, slow controlled absorption, constant plasma concentration which is maintained for a longer duration, no patient dependence for drug doses, no gastric discomfort, and flexibility of terminating the drug administration by simply removing the patch from the skin.

Rarionale of the study:The three characteristics of the pain that occurs after routine tooth extraction:(1) The Pain is usually not severe and can be managed in most patients with over-the-counter analgesics, (2) the peak pain experience occurs about 12 hours after the extraction and diminishes rapidly after that, and (3) significant pain from extraction rarely persists longer than 2 days after surgery. Non steroidal anti inflammatory drugs (ibuprofen, paracetamol etc )has the ability to reduce both pain and inflammation as a result they are the ideal analgesic agents for the control of pain in the events of surgical removal of mandibular third molar. NASIDS drugs can be administered in a variety of routes, including oral, par enteral, inhalation as well as trans dermal. Oral route is the most common for the drugs delivery. Oral NSAID may causes nephrotoxicity and hepatotoxicity'.Oral route carries the risk of first pass metabolism and loss of substantial quantities of the drug before it is absorbed systemically. Par enteral administration of drugs can be extremely painful and sudden increase in drug concentration in the plasma could lead to certain adverse effects. Trans dermal patches offer several advantages over the oral route such as bypassing first pass metabolism, slow controlled absorption, constant plasma concentration which is maintained for a longer duration, no patient dependence for drug doses, no gastric discomfort, and flexibility of terminating the drug administration by simply removing the patch from the skin. Plasma concentration of a topically applied NSAID was found to reach only a fractional level (less than 5%) of that achieved after oral administration.[8] A lower plasma drug concentration limits the systemic side effects and has an auxiliary advantage of improved action at the site of inflammation. Trans dermal delivery is associated with a lesser incidence of GI adverse effects and is particularly useful in patients unable to tolerate an oral route. However, no such reduction was documented with occurrences of heart and renal failure, which have been connected to oral NSAID usage.This study attempts to compare effectiveness of trans dermal diclofenac and oral paracetamol + ibuprofen in postoperative pain management following surgical extraction of mandibular third molar.

Sampling Method: purposive sampling

Expected sample size: study will be carried in 108 people visiting in oral and maxillofacial department, BPKIHS for surgical extraction of mandibular third molar.

Procedure: All consecutive participants who met the inclusion criteria will allocated to the oral paracetamol-500mg and ibuprofen-400mg ( group A) or trans dermal diclofenac-200mg ( group B) by computer generated random number .The surgical procedure will performed by same surgeon under same environmen using standard surgical protocol. Local anaesthesia will be provided by technique of regional blockade of the inferior and lingual alveolar nerves, with supplementary buccal nerve infiltration. A careful and slow injection of the solution will conducted after negative aspiration, with 2% lidocaine and 1:200,000 epinephrine. The incision will be given as per wards incision technique. Howarth's periosteal elevator will be used to reflect a full thickness mucoperiosteal flap and will be retracted with Austins re tractor. Buccal and distal bone removal will be done with a round bur on a straight hand piece under constant irrigation with 0.9% sterile normal saline solution and guttering done a little beyond bifurcation. After the tooth delivery socket will be inspected, irrigated and flap sutured with a 3-0 (vicryl). One suture will place just distal to the lower second molar and another on the distal aspect of the extraction socket. Duration of surgical procedure will be recorded. The post extraction instruction will be given carefully. Following removal of the impacted mandibular third molar, the oral group will given 500mg paracetamol and 400mgtablet thrice daily 30 minute while the trans dermal diclofenac group will be given diclofenac patch 200mg immediately after surgery daily for three consecutive days. Diclofenac trans dermal patch will be placed on right arm. Information on regimen and application of oral and trans dermal diclofenac was obtained from previous study[3] Patients were instructed to apply 0.12% chlorhexidine digluconate aqueous solution to control dental plaque from the second day, every 12 hours for 7 days. All patients will be given amoxicillin trihydrate. 500mg 8 hourly or erythromycin250mg 6 hourly for those who were allergic to penicillin, metronidazole 400mg 8 hourly, both for five days .pentaprazole 40 mg daily for 5 days will be given. These drugs were commenced immediately after surgery. Tramadol tablets 50mg every 8 hours will be prescribed as rescue analgesic and patients will be instructed to take it only if pain score greater than 7. consent will be taken from All subjects verbal and written patients will be taken , participaints will instructed to present to the emergency department in the event of delayed post extraction complications like uncontrolled bleeding and unbearable pain. The patients will be evaluated by the same observer. Pain will be evaluated using a Numeric Rating Scale (NRS) by telephonic interview. The assessment of pain will be done at three time points: 12, 24 and 72 hours post-operatively. The number of paracetamol tablets taken after surgery by the patients will be recorded after 3 days post -operatively.

Statistical methods proposed:

Descriptive Analysis:

Descriptive statistics, such as mean, standard deviation, median, and percentage will be applied.

Inferential statistics:

Student's t test or Mann Whitney u test will be applied to compare the observation between the two groups.

Likewise chi square test will be used to compare the proportions between two groups.

ELIGIBILITY:
Inclusion Criteria:Patients of ASA I and ASA II, who are consenting for the study.

Patient indicated for surgical extraction of mandibular third molar -

Exclusion Criteria:Hypersensitivity to local anesthetic agent Patient who are physically and mentally healthy Patient not consenting to participate in the study Pregnant females in their first and third trimester of pregnancy. Patients allergic to diclofenac and oral combination of Paracetamol and Ibuprofen.

Patient taking any analgesic at the time of surgery. Patient on anticoagulant therapy. Patient under Corticosteroids therapy. Patient needing pre-operative antibiotics prophylaxis Patient having peptic ulcerative disease. Patient having acute localized infection like pericoronitis.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
To compare the analgesic effectiveness of diclofenac trans dermal patch (200mg) and oral combination of paracetamol (500mg) and ibuprofen (400mg) following surgical removal of mandibular third molar. | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Niroj khanal, Dharān, Koshi, Nepal